CLINICAL TRIAL: NCT01510041
Title: Effects of Respiratory Muscle Training and Respiratory Exercise in Exercise Tolerance, Performing Daily Life Activities and Quality of Life of Patients With COPD.
Brief Title: Effects of Respiratory Muscle Training and Respiratory Exercise in Exercise Tolerance, Performing Daily Life Activities and Quality of Life of Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Renata Pedrolongo Basso, Principal Investigator, Master Degree, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBV-123-ER
Record Dates: First submitted 2012-01-10; First posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Physical therapy; Dyspnea; Inspiratory muscle training; Activities of daily living
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory muscle training group (Experimental)
  Interventions: Other: Inspiratory muscle training
- Respiratory exercise group (Experimental)
  Interventions: Other: Respiratory exercise

INTERVENTIONS:
Other: Inspiratory muscle training — A group will be associated with inspiratory muscle training (GTMI). The inspiratory muscle strength training will be done in the POWERbreathe ®, and the patient will breathe for two minutes, seven times with one minute rest between them, with 15% MIP, the first week, then, increased 5-10% to reach 60% of the initial MIP after four weeks. After the first month, every fifteen days the charge will be adjusted to 60% of the new value of MIP. The breathing pattern will remain free
  Arms: Inspiratory muscle training group
Other: Respiratory exercise — Specific exercise program for mobility and biomechanics of the rib cage, as exercises of the trunk and upper limbs, and stretching of large muscle groups of the trunk.
  Arms: Respiratory exercise group

SUMMARY:
In patients with chronic obstructive pulmonary disease (COPD) breaths at an abnormally high lung volume causes the inspiratory muscle to operate at non-optimal lengths, which reduce their maximal contractile forces. In addition, causes non thoraco abdominal synchronize, reduced inspiratory muscle strength and is associated with dyspnea and decreased exercise capacity. For these patients inspiratory muscle training (IMT) is a widely employed form of rehabilitation also targeting the respiratory muscle. In addition, patients often experience shortness of breath and a decline in exercise tolerance, resulting in disability in the performance of activities of daily living (ADL). The aims of this trial are to evaluate the effects of inspiratory muscle training associated with aerobic training on strength and endurance of inspiratory muscle, thoracic abdominal synchrony, exercise tolerance and quality of life patients with COPD. To compare the responses with the effects of aerobic training plus exercises of the trunk and upper limbs, and stretching of large muscle groups of the trunk. To compare difference in the perception of dyspnea during the ADL set (Borg Scale) with perception of dyspnea self-reported in the Medical Research Council (MRC), the London Chest Activity of Daily Living (LCADL) and the Pulmonary Functional Status and Dyspnea Questionnaire - Modified version (PFSDQ-M) before start the protocol. To investigate changes on perception of dyspnea (Borg scale), metabolic and ventilatory responses during a standard set of ADL tasks after a physical training and to evaluate and compare changes on perception of dyspnea. The hypothesis are that the ventilatory efficiency during the performance of ADL and the dyspnea reported from borg scale, the LCADL and the PFSDQ-M that quantifies the functional performance (change in activity levels) are improved during the IMT in conjunction with general exercise training in patients with COPD. The MIT increases the strength and endurance of inspiratory muscle, the exercise capacity and the quality of life compared to the general physical training. However, compared to the thorax abdominal synchronizes, higher modification is verified in the general physical training group with specific exercise to torso, limbs and stretching of the higher muscle group.

DETAILED DESCRIPTION:
Methodology Sample Is a prospective longitudinal. Forty patients with COPD to moderate to very severe obstruction (ratio [FEV1/FVC] <70%) and FEV1 <80% predicted (RABE et al., 2008), age ranging from 50 to 80 years old, both sexes will be assessed and treated. All subjects carry out spirometry before and after bronchodilator (BD) under medical supervision.

Experimental Procedure Patients with COPD will undergo a physical assessment of general and specific respiratory system and receive guidance on the tests and treatments proposed in this study. All of them will be instructed to maintain the medication prescribed.

The evaluation will include the following tests: medical history, St George's Respiratory Questionnaire, Medical Research Council (MRC), assessing the strength and endurance of respiratory muscle, spirometry, maximal exercise testing endurance test of the lower limbs, the Six Minute Walk Test and plethysmography of inductance.

Assessment of respiratory muscle strength The assessment of respiratory muscle strength will consist of measures of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), performed according to Black and Hyatt (1969). The measures will be carried out using a manometer scaled in cmH2O (Ger-Ar) fitted with an adapter nozzle, which contains a hole two millimeters in diameter to eliminate the pressures of facial muscles. The subjects carry out the measures in standing posture using a nose clip. The MIP will be measured by a maximal inspiration, preceded by a maximal expiration starting from residual volume, and MEP will be measured by a maximal expiration, preceded by a maximal inspiration based on the total lung capacity. The inspiratory and expiratory must be maintained for at least one second. Will be performed at least three and maximum five measures will be considered acceptable if there is a difference of 10% or less between them. The highest value will be used for statistical analysis. The patients will be allowed a one-minute rest between measurements.

Assessment of respiratory muscle endurance Incremental and constant tests After measurements of MIP the endurance of the inspiratory muscles using the PowerBreathe® will be evaluate.

The test starts with incremental 10cmH2O (which is the minimum load of the unit) and every two minutes there will be an increase 10cmH2O, and conducted a further minute before increasing the load. The biggest load you can sustain for at least one minute is the maximum that will be considered. The test will be held constant at 80% of the pressure in the incremental test, to determine the time limit for implementation, considering 30 minutes as the maximum time (FIZ et al., 1998; RAMIREZ-SARMIENTO et al., 2002).

In both tests the breathing pattern will be free and the breathing frequency will be noted. Besides the pressure generated will be monitored by a manometer attached to PowerBreathe® .

Six Minute Walk Test (6MWT) 6MWT will be performed on a track 30 meters long and 1.5 wide, with markings every 2 feet. Tests will be conducted in accordance with the standards of the ATS (2002). Every two minutes will be checked the oxygen saturation (SpO2), heart rate (HR), the sensation of dyspnea and fatigue of the lower limbs by Borg CR10 scale. These measures associated with the measurement of blood pressure (BP) will be checked before, immediately after the test and after six minutes. It will be two tests on the same day, at intervals of 30 minutes, to avoid the effect of learning on test performance. It will be considered the greatest distance for statistical analysis.

Maximum Exercise Testing To perform this test will be followed by the Standardization of techniques and equipment for exams exercise testing and spirometry (2003), and will be conducted in a room properly heated, keeping the temperature around 18 ° C and 22 ° C and relative humidity air between 50% and 70%.

It will be performed by a cardiologist on a treadmill using modified Bruce protocol, which is a good option for those patients with low functional capacity, such as the elderly and people with respiratory and cardiovascular disease. This is a protocol in which both the speed and the incline of the treadmill are increased every three minutes and modified. The two earlier stages have lower velocities and inclination (SAMORA e VERSIANI, 2008; NEDER e NERY, 2003).

In addition, to monitoring the continuous ECG tracing at rest and at each stage are checked the values of SpO2, dyspnea and fatigue of the lower limbs by Borg CR10 scale and BP.

The criteria for interrupting the test are: elevated blood pressure (DBP) to 120 mmHg, sustained drop in systolic blood pressure (SBP), marked elevation of SBP 260mmHg up, reaching the maximum HR (HRmax) provided by age, fall in SpO2 below 80%, ECG abnormalities, the patient's request due to physical exhaustion, dyspnea disproportionate to the exercise intensity, pain in lower limbs, dizziness or chest discomfort; failure of monitoring systems and / or record.

Test of endurance of the lower limbs This test will be conducted on a treadmill for up to 30 minutes at an intensity of 80% of the speed and slope obtained at maximal exercise testing.

Inductance plethysmography For this test it will use a system of respiratory inductive plethysmography (LifeShirt; Vivo Metrics; Ventura, CA), whose sensors are two electrical conductors sewn to a sleeveless vest, and stay in the region of the nipples and the umbilical region. There are three electrodes placed in predetermined areas and connected for a portable, battery, which records the SpO2, electrocardiogram (ECG) and body movements in three axes (CLARENBACH et al., 2005).

This is a highly reliable instrument used to monitor the volume and time components of breathing pattern and thoracoabdominal configuration. It is based on changes in cross-sectional area that occur in the compartments of the chest and abdomen. The method is minimally invasive, requires no mouthpiece or nose clip (except for calibration), and there is therefore need for direct contact with air. The accuracy of plethysmography to provide tidal volume values is satisfactory and depends on an initial calibration and proper maintenance of the same body position. The equipment will be calibrated in advance the measures according to the instructions of the device in all subjects. In this study, the following variables will be analyzed by plethysmography, tidal volume (Vt), respiratory rate (RR), minute ventilation (VE), the ratio between time to reach peak inspiratory flow and inspiratory time (PIFT / Ti), flow mean inspiratory (Vt/Ti), percent rib cage contribution to tidal volume (%RC/Vt) and phase angle (PhAng) (CLARENBACH et al., 2005; PARREIRA et al, 2005).

These measures will be carried out at 90 degrees sitting and standing, resting and doing exercises with their arms, and walking, to see whether dyssynchrony occurs. The signal acquisition will total duration of 30 minutes.

Perception of dyspnea assessed by different scales and questionnaires. It will perform a set of ADL tasks (making bed, taking shower, putting on clothes, brushing teeth and combing hair, lifting containers on a shelf at eye level and lifting and lowering containers on a shelf above the scapular waist) patients will evaluate by Borg scale for dyspnea and a portable system will be used to assess ventilator parameters, oxygen consumption, carbon dioxide production and heart rate during standardized: wake up and making bed, taking shower and washing one's back, putting on clothes, brushing teeth and combing hair, lifting and lowering containers on a shelf at eye level, lifting and lowering containers on a shelf above the scapular waist and hanging. No specific amount of time is stipulated; the patient is only instructed to complete the task. During the set of ADL a metabolic system (MedGraphics VO2000 St. Paul MN, USA) is used. In addition, these patients will self-report the MRC, LCADL scale and PFSDQ-M, before the start of the protocol to investigate the difference and the correlation between these instruments.

Training Program After testing and pre-experimental tests, subjects will be randomly divided into two groups. The treatment program will consist of sessions with duration of about 1 hour or 1 hour and 30 minutes depending on the training, three times per week on alternate days for 16 consecutive weeks, totaling 48 sessions.

Before the beginning and end of the sessions will be verified measures of blood pressure (BP), SpO2, HR. Measures of HR, SpO2 and BP will be obtained during the session for monitoring.

All patients will undergo a general physical training. In this training will be conducted stretches of upper and lower limbs, treadmill exercise with HR between 70-80% HR max obtained at maximum exercise test, which could be carried out continuously or with intervals, up to a maximum of 30 minutes, and resistance exercises to LL, using free weights, with progressive increases of ½ kg each month to reach 2 kg in the last month.

A group will be associated with inspiratory muscle training (GTMI). The inspiratory muscle strength training will be done in the POWERbreathe ®, and the patient will breathe for two minutes, seven times with one minute rest between them, with 15% MIP, the first week, then, increased 5-10% to reach 60% of the initial MIP after four weeks. After the first month, every fifteen days the charge will be adjusted to 60% of the new value of MIP. The breathing pattern will remain free, but the patient will be instructed to release all the air, not to hyperventilate (HILL et al, 2007).

In other group of patients will be associated a specific exercise program for mobility and biomechanics of the rib cage, called respiratory exercise group (GCR), as exercises of the trunk and upper limbs, and stretching of large muscle groups of the trunk.

Upon completion of the protocol will all be assessed.

ELIGIBILITY:
Inclusion Criteria:

* the patients with clinical diagnosis of COPD presenting FEV1/FVC < 70% and FEV1 < 80% predicted by pulmonary function observed and were classified as patients with moderate to very severe obstruction (RABE et al., 2008),
* clinically stable with no history infection or exacerbation of the respiratory symptoms or
* a change in medication for two months preceding the study.
* the patients were non oxygen dependent, smokers or former smokers.

Exclusion Criteria:

* patients with clinical diagnosis of COPD presenting FEV1/FVC ≥ 70% FEV1 ≥ 80% predicted (RABE et al., 2008)
* who present respiratory, cardiac, rheumatic, musculoskeletal, orthopedic and neuromuscular disorders associated that may prevent them of the testing and intervention proposed,
* that are experiencing swelling in lower limbs,
* that change the type of medication during the study,
* uncontrolled hypertension patients,
* saturation below 90% at rest and
* did not agree to sign the formal consent form proposed.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Renata P Basso, Ms, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of Sao Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Fiz JA, Romero P, Gomez R, Hernandez MC, Ruiz J, Izquierdo J, Coll R, Morera J. Indices of respiratory muscle endurance in healthy subjects. Respiration. 1998;65(1):21-7. doi: 10.1159/000029223. PMID 9523364
- [Background] Ramirez-Sarmiento A, Orozco-Levi M, Guell R, Barreiro E, Hernandez N, Mota S, Sangenis M, Broquetas JM, Casan P, Gea J. Inspiratory muscle training in patients with chronic obstructive pulmonary disease: structural adaptation and physiologic outcomes. Am J Respir Crit Care Med. 2002 Dec 1;166(11):1491-7. doi: 10.1164/rccm.200202-075OC. Epub 2002 Jul 19. PMID 12406842
- [Background] Samora GAR, Versiani LC. Diretrizes básicas da fisiologia do exercício para avaliação da capacidade funcional. In: Machado MGR. Bases da fisioterapia respiratória. Terapia intensiva e reabilitação. 1ª Edição, Rio de Janeiro, Guanabara-Koogan, 2008.
- [Background] Clarenbach CF, Senn O, Brack T, Kohler M, Bloch KE. Monitoring of ventilation during exercise by a portable respiratory inductive plethysmograph. Chest. 2005 Sep;128(3):1282-90. doi: 10.1378/chest.128.3.1282. PMID 16162719
- [Background] Parreira VF, Tomich GM, Britto RR, Sampaio RF. Assessment of tidal volume and thoracoabdominal motion using volume and flow-oriented incentive spirometers in healthy subjects. Braz J Med Biol Res. 2005 Jul;38(7):1105-12. doi: 10.1590/s0100-879x2005000700014. Epub 2005 Jul 4. PMID 16007282
- [Background] Hill K, Jenkins SC, Philippe DL, Shepherd KL, Hillman DR, Eastwood PR. Comparison of incremental and constant load tests of inspiratory muscle endurance in COPD. Eur Respir J. 2007 Sep;30(3):479-86. doi: 10.1183/09031936.00095406. Epub 2007 May 15. PMID 17504795
- [Background] Neder JR, Nery LE. Fisiologia Clínica do Exercício. 1ª Edição, São Paulo, Artes Médicas, 2003.
- [Background] Sociedade Brasileira de Cardiologia. [Standardization of techniques and devices for ergometric and ergospirometric exams]. Arq Bras Cardiol. 2003 Apr;80(4):457-64. Epub 2003 Apr 29. No abstract available. Portuguese. PMID 12754567
- [Derived] Basso-Vanelli RP, Di Lorenzo VA, Labadessa IG, Regueiro EM, Jamami M, Gomes EL, Costa D. Effects of Inspiratory Muscle Training and Calisthenics-and-Breathing Exercises in COPD With and Without Respiratory Muscle Weakness. Respir Care. 2016 Jan;61(1):50-60. doi: 10.4187/respcare.03947. Epub 2015 Nov 10. PMID 26556894